CLINICAL TRIAL: NCT00787371
Title: Study to Confirm Dose Response With PegIntron (SCH 54031) Monotherapy in Patients With Chronic Hepatitis C
Brief Title: Effect of Low-dose PegIntron on ALT Normalization in Japanese Patients With Chronic Hepatitis C (Study P04508)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04508; JPC-04-356-20
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
Keywords: alanine transaminase
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.25 Dose Group (Experimental): PegIntron 0.25 mcg/kg SC QW for 12 weeks
  Interventions: Biological: PegIntron (peginterferon alfa-2b)
- 0.5 Dose Group (Experimental): PegIntron 0.5 mcg/kg SC QW for 12 weeks
  Interventions: Biological: PegIntron (peginterferon alfa-2b)
- 1.0 Dose Group (Experimental): PegIntron 1.0 mcg/kg SC QW for 12 weeks
  Interventions: Biological: PegIntron (peginterferon alfa-2b)
- No-treatment Control (No Intervention): No treatment (no placebo)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b) — PegIntron 0.25 mcg/kg subcutaneously (SC) once a week (QW) for 12 weeks
  Other Names: PegIntron, peginterferon alfa-2b, SCH 54031
  Arms: 0.25 Dose Group
Biological: PegIntron (peginterferon alfa-2b) — PegIntron 0.5 mcg/kg SC QW for 12 weeks
  Other Names: PegIntron, peginterferon alfa-2b, SCH 54031
  Arms: 0.5 Dose Group
Biological: PegIntron (peginterferon alfa-2b) — PegIntron 1.0 mcg/kg subcutaneously (SC) once a week (QW) for 12 weeks
  Other Names: PegIntron, peginterferon alfa-2b, SCH 54031
  Arms: 1.0 Dose Group

SUMMARY:
In patients with chronic hepatitis C, the ultimate treatment goal is the improvement of liver histology and inhibition of progression to liver cirrhosis and hepatocellular carcinoma (HCC). These effects are reported to be correlated with sustained ALT improvement. Therefore, the aim of this study is to determine if a low-dose (0.25, 0.5, or 1.0 mcg/kg SC QW) PegIntron monotherapy administered for 12 weeks will result in ALT normalization in Japanese patients with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic hepatitis C patients (CHC) who met all of the following criteria:

* At least 20 years of age and willing to sign an informed consent
* Patients who can practice contraception
* Patients who are classified either as relapsers or non-responders.
* Weight between 45 and 100 kg
* Patients willing to be hospitalized for 3 days after the start of treatment
* Patients with positive HCV-RNA
* Serum ALT level: Over 60 IU/L, equal to or less than 150 IU/L
* Neutrophil count: equal to or more than 1,200 /mm^3
* Platelet count：equal to or more than 100,000/mm^3

Exclusion Criteria:

* Patients with conditions which would interfere with the evaluation of therapeutic efficacy of the study drug and patients for whom assurance of safety is a concern were excluded from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who achieve normalization of ALT in each treatment group | Measured at the end of 12 weeks of treatment or at discontinuation.

SECONDARY OUTCOMES:
Safety: adverse events, adverse reactions, laboratory test result (hematology, blood biochemistry and thyroid function test) | Measured between when the patient signs the informed consent form and the end of post-treatment follow-up

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html